CLINICAL TRIAL: NCT04786314
Title: The Effect of Hot and Cold Water Application to Pregnant Women With Restless Legs Syndrome on Complaints and Quality of Sleep
Brief Title: The Effect of Hot and Cold Water Application on Pregnant Women With Restless Leg Syndrome
Acronym: RLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ozlem Kaplan, Reserch Asistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TDK-2020-10628
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Restless Legs Syndrome; Pregnant; Sleep Disorder
Keywords: Restless legs syndrome; Pregnant; Cold Water Application; Hot Water Application; Quality of Sleep
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hot Water Application Group (Experimental): Pregnant women will apply hot water to their legs before going to sleep for a week, depending on the groups they are in.
  Interventions: Other: Hot Water Application
- Cold Water Application Group (Experimental): Pregnant women will apply cold water to their legs before going to sleep for a week, depending on the groups they are in.
  Interventions: Other: Cold Water Application
- Control Group (No Intervention): There will be no intervention other than routine follow-up and maintenance.

INTERVENTIONS:
Other: Hot Water Application — Pregnant women will apply hot water to their legs before going to sleep for a week.
  Arms: Hot Water Application Group
Other: Cold Water Application — Pregnant women will apply cold water to their legs before going to sleep for a week.
  Arms: Cold Water Application Group

SUMMARY:
This study was planned as a randomized controlled study to determine the effect of hot and cold water application on complaints and sleep quality in pregnant women with restless legs syndrome (RLS). Pregnant women with a total of 90 RLS, including 30 people in each group, will be included in the study. The data of this study will be collected by Personal Information Form, RLS Diagnosis Criteria Questionnaire, RLS Severity Rating Scale, Pittsburgh Sleep Quality Index, Post Application Follow-up Chart and Application Satisfaction Form.

While hot and cold water is applied in the intervention groups in the study, no application other than routine maintenance and follow-up will be done to the control group.Data analysis obtained in the research will be performed in TURCOSA statistical software (Turcosa Analytics Ltd Co, Turkey, www.turcosa.com.tr).In comparisons, a value of p <0.05 will be considered statistically significant.In order to conduct the study, the necessary Academic Committee decision, Ethics Committee approval (September 09, 2020 and number 2020/445) and institutional permission were obtained. The individuals included in the study will be informed about the purpose of the research, their verbal consent will be obtained and the participant's informed consent form will be signed.

ELIGIBILITY:
Inclusion Criteria:

1. Least literate
2. 24-32. between the weeks of gestation
3. Having a single pregnancy
4. The presence of RLS is detected according to the RLS Diagnostic Criteria Questionnaire
5. Having RLS due to pregnancy
6. Uses Iron, Vitamin D, Magnesium and Calcium
7. Pregnant women who have a severity of 11 or more according to the RLS Severity Rating Scale will be included in the study

Exclusion Criteria:

1. Those who have a communication disability,
2. Risky pregnancy (Preterm labor risk, Cervical insufficiency, etc.),
3. Chronic disease (Diabetes, Hypertension, Thyroid, Cardiovascular disease, epilepsy, etc.),
4. With maternal obesity, BMI> 30
5. He has heirs in his legs,
6. Pre-pregnancy sleep apnea,
7. Having any psychiatric disease and using antipsychotic, antidepressant medication,
8. Using antihistamine, antiepileptic, antiemetic, calcium channel blocker, dextromethorphan and decongestant type drugs,
9. Using heparin,
10. Pregnant women with a history of deep vein thrombosis, or atherosclerosis history or risk will not be included in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Since the study will be conducted with pregnant women with restless legs syndrome, only women were included in the study.
Enrollment: 90 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
RLS Severity Rating Scale | change from baseline score at the end of one week
  The RLS Severity Rating Scale was developed in 2003 by the International Restless Legs Syndrome Study Group. The scale was applied in the selection of patients and in the weekly evaluation of RLS severity. The scale comprised ten questions; each question was scored between 0 and 4. Questions 1, 2, 4, 6, 7, and 8 were related to RLS symptoms, questions 5, 9, and 10 were related to the effect of the disease on the mental state and daily social activities of patients with RLS, and question 3 was about the diagnostic criteria of RLS. The overall score indicated the RLS severity. A minimum score of 0 and a maximum score of 40 could be obtained. A score between 1 and 10 corresponded to "mild," 11-20 "moderate," 21-30 "severe," and 31-40 "very severe" RLS.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | change from baseline score at the end of one week
  The form consists of a total of 24 questions. Each question is scored between 0 and 3. Pittsburgh Sleep Quality Index score in the 0-21 range, with high scores indicating poor sleep quality. If the Pittsburgh Sleep Quality Index global score is greater than 5, it indicates that the sleep quality is significantly worse. The fact that the Pittsburgh Sleep Quality Index score is above 5 indicates that the person has serious trouble in at least two areas related to his sleep, or that he has mild or moderate difficulty in more than three areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will be shared after the study ends.